CLINICAL TRIAL: NCT00535704
Title: Preventing Substance Use and Risky Behavior Among Rural African American Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01DA021736-01 (NIH)
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2014-04

CONDITIONS: Risky Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): The Strong AFrican American FAmilies-Teen program is a five part educational program has been designed to help teens and their parents create successful futures and avoid the risky behaviors that sometimes keep teens from reaching their goals.
  Interventions: Behavioral: Strong African American Families-Teen Program
- 2 (Other): The FUEL program is a family-based adaptation of a curriculum designed to assist teens to develop lifestyles that prevent health problems such as heart disease, diabetes, and being overweight. This program deals with diet and exercise, the influence of TV and magazines on eating habits, and handling stress.
  Interventions: Behavioral: FUEL

INTERVENTIONS:
Behavioral: Strong African American Families-Teen Program — 5 week educational program for teens and their caregivers.Each meeting lasts approximately 2 hours.
  Arms: 1
Behavioral: FUEL — 5 week educational program for teens and caregivers. Each weekly session lasts approximately 2 hours
  Arms: 2

SUMMARY:
The Rural African American Families Health (RAAFH) Project is a federally funded research study designed to evaluate the effectiveness two prevention programs designed for rural African American families. One program, FUEL, helps teens develop lifestyles that prevent health problems such as heart disease, diabetes, and being overweight. This program deals with diet and exercise, the influence of TV and magazines on eating habits, and handling stress. The second program, the Strong African American Families Teen Program (SAAF-T), helps teens learn how to develop plans for the future and to avoid drug use and unsafe sex. The sessions deal with goal setting, peer pressure, and staying in school.

ELIGIBILITY:
Inclusion Criteria:

* African American student in 10th grade
* Agree to randomization and assessment
* Resides in targeted county
* Target and parent speak English

Exclusion Criteria:

* Active psychoses

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 502 (Actual)
Dates: Start 2007-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Sexual behavior | 3 months

SECONDARY OUTCOMES:
Substance Use | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gene H Brody, Principal Investigator — University of Georgia
Locations (1):
- Center for Family Research, Athens, Georgia, United States